CLINICAL TRIAL: NCT00075933
Title: A Phase I Clinical, Pharmacokinetic Study of ARQ 501 in Subjects With Advanced Solid Tumors
Brief Title: ARQ 501 in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 501-101
Record Dates: First submitted 2004-01-12; First posted 2004-01-13 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — beta-lapachone

INTERVENTIONS:
Drug: ARQ 501

SUMMARY:
ARQ 501, an investigational anticancer drug, is intended to selectively kill cancer cells and spare normal cells by restoring and activating cellular checkpoints known to be defective in cancer using the Company's unique biology platform, Activated Checkpoint Therapy™ (ACT).

ARQ 501 has the potential for improved activity and reduced toxicity over other molecular approaches and traditional cancer chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed solid tumor that is metastatic, unresectable or recurrent and for which standard curative or palliative measures do not exist or are no longer effective.
* ECOG performance status greater than or equal to 1
* Life expectancy greater than three months
* Acceptable pretreatment clinical laboratory results

Exclusion Criteria

* Subjects who have had chemotherapy or radiotherapy within 4 weeks
* Subjects receiving any other investigational agents
* Subjects with known untreated brain metastases
* Subjects receiving hepatic enzyme-inducing antiseizure drugs ("EIASD")
* Subjects with uncontrolled intercurrent illnesses
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey I Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute; C. Casey Cunningham, MD, Principal Investigator — Mary Crowley Medical Research Center
Locations (2):
- United States (2):
  - Dana Farber/Partners CancerCare Inc, Boston, Massachusetts
  - Mary Crowley Medical Research Center, Dallas, Texas